CLINICAL TRIAL: NCT02878304
Title: Recovery of Hand Function After Stroke- a Longitudinal Study Using Novel Methods to Quantify Hand Function and Connectivity in Brain Networks
Brief Title: Biomarkers for Prediction of Hand Function After Stroke - The ProHand Study
Acronym: ProHand
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danderyd Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROHAND_001
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Hemiparesis
Keywords: Prognosis; Hand function; Rehabilitation; Spasticity; MRI
MeSH Terms: conditions — Stroke; Paresis; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall aim is to identify key determinants for recovery of hand function after stroke by applying newly developed hand function measures together with MRI measurements of the lesioned cerebral structures.

DETAILED DESCRIPTION:
Almost half of surviving stroke patients are left with impaired function of the hand but individual profiles of weakness, spasticity, sensory and bimanual function vary widely. Improved prediction of recovery after stroke has broad implications for clinical decisions on the type, duration and goals of rehabilitation.

100 consecutive patients with 1st ever stroke and upper limb hemi-paresis will be subject to imaging, at 4 weeks and 6 months, and behavioral assessments at 4 weeks, 3 months and 6 months after stroke. The imaging protocol includes anatomical sequences for lesion mapping, diffusion tensor imaging and resting-state functional MRI for structural and functional connectivity analyses, respectively. Clinical hand function measures will be combined with novel validated methods to quantify spasticity,grip force control, sensory and bimanual function.

ProHand will provide insights into neural mechanisms related to recovery of hand function after stroke and enable enhanced prediction and development of targeted treatment trials.

ELIGIBILITY:
Inclusion Criteria:

* first ever stroke and clinically diagnosed arm paresis

Exclusion Criteria:

* incapability to give informed concent and/or understand and comply with instructions, other disorders that may affect hand function (e.g. other neurological conditions, arthritis), cerebellar lesions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited at entry to a specialized sub-acute rehabilitation unit after first time stroke
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment for Upper Extremity | From 4 weeks to 3 and six months

OTHER OUTCOMES:
Structural and functional connectivity measures; functional Magnetic Resonance Imaging | From 4 weeks to 6 months
Change in NeuroFlexor(C) measures | From 4 weeks to 3 and 6 months
  Quantitative measures of the neural and biomechanical components of the force resisting passive movement of ther wrist
Change in modulation of gripforce: Visuomotor grip force tracking task | From 4 weeks to 3 and 6 months
Change in Action Research Arm Test, ARAT | From 4 weeks to 3 and 6 months
Change in Strength-Dexterity test | From 4 weeks to 3 and 6 months
  Dexterous ability/quantification of precision in finger movements
Change in grip force | From 4 weeks to 3 and 6 months
  Dynamometry
Change in Assisting Hand Assessment, AHA | From 4 weeks to 3 and 6 months
  Measures of the spontaneous use of the more affected hand in specific bimanual activities
Change in Box and Block Task, BBT | From 4 weeks to 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jörgen Borg, Professor, Study Director — Department of Rehabilitation Medicine, Danderyd University Hospital, Karolinska Institutet
Locations (1):
- Danderyd University Hospital, Stockholm, Danderyd, Sweden

REFERENCES:
- [Derived] Plantin J, Verneau M, Godbolt AK, Pennati GV, Laurencikas E, Johansson B, Krumlinde-Sundholm L, Baron JC, Borg J, Lindberg PG. Recovery and Prediction of Bimanual Hand Use After Stroke. Neurology. 2021 Aug 17;97(7):e706-e719. doi: 10.1212/WNL.0000000000012366. Epub 2021 Jun 14. PMID 34400568
- [Derived] Hybbinette H, Ostberg P, Schalling E. Intra- and Interjudge Reliability of the Apraxia of Speech Rating Scale in Early Stroke Patients. J Commun Disord. 2021 Jan-Feb;89:106076. doi: 10.1016/j.jcomdis.2020.106076. Epub 2021 Jan 6. PMID 33493822
- [Derived] Pennati GV, Plantin J, Carment L, Roca P, Baron JC, Pavlova E, Borg J, Lindberg PG. Recovery and Prediction of Dynamic Precision Grip Force Control After Stroke. Stroke. 2020 Mar;51(3):944-951. doi: 10.1161/STROKEAHA.119.026205. Epub 2020 Jan 7. PMID 31906829